CLINICAL TRIAL: NCT06905626
Title: Prevention of Obesity in Adolescents and Young Adults
Brief Title: Weight Gain Prevention in Adolescents and Young Adults
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEDS-2024-33047
Record Dates: First submitted 2025-02-04; First posted 2025-04-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Obesity prevention
MeSH Terms: interventions — Qsymia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study will have a 1:1 randomization. Participants will receive either Qsymia or a matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qsymia arm (Experimental): Qsymia
  Interventions: Drug: Qsymia 7.5 miligrams (mg)-46 mg Extended Release Capsule
- Placebo arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qsymia 7.5 miligrams (mg)-46 mg Extended Release Capsule — Qsymia
  Other Names: Qsymia
  Arms: Qsymia arm
Drug: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
The investigators believe they key to effective prevention of obesity is early identification of individuals at high risk of excess weight gain and proactive implementation of a comprehensive approach including lifestyle-based coaching and preventive medical management targeting the pathophysiology of dysregulated energy metabolism. In this study the investigators will take a fundamentally different approach to the science of obesity prevention by targeting the underlying biological processes driving unhealthy weight gain in adolescents/young adults (AYAs), a group that has been underrepresented in medication trials.

DETAILED DESCRIPTION:
Once obesity develops and becomes entrenched, achieving sustained weight loss is extremely difficult. Thus, preventing the accumulation of excess adiposity in high-risk individuals is the ideal course of action. AYAs are high-risk individuals, as this is a life stage characterized by susceptibility for accelerated weight gain. However, most obesity prevention interventions targeting AYAs have reported null findings or modest effects. It is possible that failure to address the underlying physiology of the energy regulatory system is at least partly responsible for the underwhelming results. Numerous physiological mechanisms drive weight gain by stimulating appetite and food palatability, as well as influence other weight related behaviors to achieve a predetermined body weight set point. Previous obesity prevention interventions in AYAs have almost entirely focused on modifying individual behaviors and/or external environmental conditions and have not addressed the biological pathways driving energy regulation. Effectively targeting the underlying physiological processes promoting body fat storage, such as with pharmacotherapy, may be an essential component of successful obesity prevention for some individuals.

When used in combination with lifestyle-based weight gain prevention counseling, low-dose preventative pharmacotherapy has the potential to halt or slow unhealthy weight gain in AYAs by targeting key mechanisms in the energy regulatory system. Qsymia is among the most cost-effective anti-obesity medications approved for adolescents and adults. Its mechanisms of action may be ideal for impeding weight gain and ultimately preventing the onset of obesity because they are multifactorial and involve reducing appetite, enhancing satiety, and potentially increasing energy expenditure. Moreover, flexible dosing with Qsymia provides the option to introduce preventative pharmacotherapy at low levels of exposure (minimizing risk) yet allows for dose escalation if weight gain were to ensue. It is also attractive in the context of prevention owing to its oral route of administration and relatively low cost compared to other medications.

In the proposed clinical trial, the investigators plan to diverge significantly from historical obesity prevention approaches by pairing lifestyle-based weight gain prevention coaching with low-dose preventative pharmacotherapy to target the underlying biological processes implicated in weight gain. The investigators will target AYAs (18 to <25 years old) at high risk of developing obesity: defined as those with a body mass index (BMI) between 25-29.9 kg/m^2 (overweight classification) and a family history of obesity (one biological parent with severe obesity and/or two biological parents with obesity). The investigators will randomize 140 of these individuals (1:1) to Qsymia or placebo with both groups additionally receiving lifestyle-based weight gain prevention coaching. Over a period of two years, the investigators will: 1) compare changes between groups in BMI trajectories as well as incidence of obesity and regression to normal weight; 2) determine if there are differences between groups in diet quality and eating behaviors; and 3) investigate changes in visceral adipose tissue and its relation to cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to M 25 at screening
* BMI >/= 25 to < 30 kg/m^2
* Family history of obesity defined as one biological parent with severe obesity (BMI >/= 35) and/or two biological parents with obesity (BMI >/=30). Parental obesity status will be confirmed by obtaining a release of information to review and electronic health record.

Exclusion Criteria:

* Tanner stage 1-4
* Diabetes (type 1 or 2)
* Current or recent (<6 months prior to screening) use of anti-obesity medication(s) or other weight-altering medication(s) (e.g. atypical anti-psychotics, attention deficit hyperactivity disorder (ADHD) stimulant)
* Previous bariatric surgery
* Current or recent (<6 months prior to screening) use of medication(s) to treat insulin resistance
* Recent initiation (<3 months prior to screening) of anti-hypertensive or lipid medication(s)
* History of glaucoma
* Current or recent (<14 days prior to screening) use of monoamine oxidase inhibitor
* Known hypersensitivity to sympathomimetic amines
* History of treatment with growth hormone
* Patient Health Questionnaire-9 (PHQ-9) score of >/= 15 at screening
* Eating disorder symptoms within 6 months and/or any past medical diagnosis of eating disorder
* Major psychiatric disorder
* Unstable clinically-diagnosed depression
* History of suicide attempt
* Suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at any time during the study
* Current pregnancy or breastfeeding
* Plans to become pregnant
* If sexually active, refusal to use 2 forms of birth control
* Tobacco use
* Alanine transaminase (ALT) or aspartate transaminase (AST) >/= 2.5 times the upper limit of normal
* Bicarbonate 18 mmol/L
* Creatinine > 1.2 mg/dL
* Creatinine clearance <50 mL/min (Schwartz formula)
* History of seizures
* Uncontrolled hypertension
* History of structural heart defect
* History of clinically significant arrhythmia
* Diagnosed monogenic obesity
* History of cholelithiasis
* History of nephrolithiasis
* Hyperthyroidism
* Untreated thyroid disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
BMI | 24 months
  Change in body mass index

SECONDARY OUTCOMES:
Diet quality and eating behaviors | 24 months
  Daily caloric intake

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Kelly, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: Yes
A long-term data sharing and preservation plan will be used to store and make publicly accessible the data beyond the life of the project. The deidentified data will be deposited into the Data Repository for University of Minnesota (DRUM). This University of Minnesota Libraries hosted institutional data repository is an open access platform for dissemination and archiving of university research data and is free to the University of Minnesota researchers. Curators review all incoming submissions and work with data authors to comply with data sharing requirements in ways that make data FAIR (Findable, Accessible, Interoperable, Reusable).
Supporting Information: Study Protocol, SAP
Time Frame: 10 years
Access Criteria: U of Minnesota Libraries